CLINICAL TRIAL: NCT06858904
Title: Rehydration With a Trace Mineral Supplement
Acronym: TRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Stavros Kavouras, Professor and Assistant Dean, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00021498
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Dehydration (Physiology)
Keywords: rehydration; sports drinks; fluid balance; water retention
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ConcenTrace (Experimental): Beverage with ConcenTrace minerals
  Interventions: Dietary Supplement: ConcenTrace
- ZeroLyte (Experimental): Beverage with high level of trace elements but no sugar
  Interventions: Dietary Supplement: ZeroLyte
- Placebo (Placebo Comparator): Water with non caloric, non-sodium containing sweetner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Non- calorically sweetened Water
  Arms: Placebo
Dietary Supplement: ConcenTrace — 1.25 milliliter of concentrace per liter
  Arms: ConcenTrace
Dietary Supplement: ZeroLyte — Beverage with 1 pack of ZeroLyte per 500 milliliter of water
  Arms: ZeroLyte

SUMMARY:
It is well established that post-exercise rehydration with electrolyte solutions is more effective than plain water. However, most commercially available drinks are high in electrolytes but lack some essential trace minerals. This study aims to examine the impact of a higher-electrolyte sports drink compared with a low-electrolyte, trace-mineral-rich solution and water on the time course and extent of rehydration after exercise-induced dehydration.

DETAILED DESCRIPTION:
Protocol Before the start of the study eligible participants will visit our lab to conduct a screening of medical history, weight, height, and a onetime assessment of body composition via BIA and Training history. This visit will take place at least one day before the actual start of the study and typically lasts no longer than 30 minutes. During this visit participants will be given two questionnaires, one regarding the physical activity readiness of the participant, and another one regarding their health history. If a participant does not meet the physical criteria and does not pass both questionnaires, they will be given a $25 digital Tango gift card for their brief visit to our lab. Participants who do pass will be given a scheduled date and time to visit the lab again for their first official trial.

At the start of the study subjects will visit the lab after at least 10h of fast and they will consume a light breakfast. An intravenous catheter will be place in an antecubital vein and a blood sample will be taken after 20 min for baseline. A baseline skin hydration reading will also be taken at this time. Subjects will void their bladders and a body weight will be taken.

Dehydration:

Consistent with the study by Shirreffs et al (2007) and based on our previous work, dehydration will be accomplished on the morning of testing via mild exercise and heat exposure to elicit a body weight loss of -2%. The subjects will perform four bouts of 25-minutes low-intensity exercise and 5 min rest (alternating cycling & walking) or till they reach -2% of body weight dehydration.

Rehydration:

Upon losing 2% body weight, participants will be instructe to rinse off their face to get rid of excess sweat. This is followed by a 20 minutes rest period in a thermo-comfortable environment, a dehydrated baseline blood sample will be taken, along with a dehydrated skin hydration reading and subject will start the rehydration protocol.

The volunteers will consume one of the three drinks below in a cross over balance mode. During the first hour four equal doses will be consumed in15-minutes intervals at a total volume of 150% of their body weight loss.

Trials/Drinks (block randomization will be used to assign individual participants to each specific trial/drink using their ID number):

* Water
* ConcenTrace®
* ZEROLyte™ Note: The beverage volumes will be standardized at 150% of body weight loss during exercise-induced dehydration to ensure consistency across trials.

See the study design expressed as a figure below:

Measurements:

All measurements will be performed at one of the test rooms at our lab facility that boarders the room where participants can relax and wait out the end of the study day. When certain measurements need to be performed they simply move from one room to the next. Duration of taking blood and urine samples will take not more than 30-90 seconds each and perceptual data will take 30-60 seconds to be reported. To allow to perform all measurements, participants will remain supervised by a team member in the lab for up to 7 hours per trial. Therefore, there will be a separate space available that allows for self-study or watching TV that includes a chair and table to work on and a couch to relax.

Blood samples (7 per trial):

Blood samples will be taken via a venous catheter attached to an extension tube and a stopcock. After each blood sample sterile saline solution will be infused in the extention tube to avoid clotting. The iv catheter will be placed by one of the Clinical Research Center phlebotomists. A total of seven 10 milliliters blood samples will be collected on the euhydrated baseline, dehydrated baseline and at 30, 60, 120, 180, and 240 minutes of the rehydration period.

All samples will be analyzed for glucose, osmolality, total plasma protein, hematocrit, hemoglobin (for plasma volume changes), sodium, potassium, and chloride.

Urine samples (6 per trial):

Urine samples will be provided from the subjects in a urine cup. The cup will be placed in the pass-through window where a lab technician will receive it and process it.

Urine samples will be collected using ~900 milliliters cups at euhydrated baseline, dehydrated baseline and cumulative totals will be collected at 60, 120, 180, and 240 minutes of the rehydration period. All samples will be analyzed for urine osmolality, specific gravity, volume, sodium, and potassium.

Sweat samples (1 per trial):

Sweat samples will be collected with sweat patches. The sweat patches are like a band-aid that it will be placed on the forearm and stay there for approximately 30 min to absorb sweat. After 30 minutes the patch will be removed and the sweat sample will be extracted by centrifugation in the lab.

Sweat samples will be collected during the first 30 min of exercise to assess sodium and potassium content.

Skin Hydration (6 per trial):

Skin hydration will be measured with a pen-like instrument that applies a very light pressure on the skin. This does not cause any pain or skin irritation.

Skin hydration will be measured on the face (inner zygomatic bone), arm (bicep brachii) at euhydrated baseline, 30 minutes after the end of dehydration, and at 60, 120, 180, and 240 minutes of rehydration.

Gastrointestinal Symptoms (6 per trial):

Gastrointestinal symptoms will be assessed at 1, 2, 3 and 4 hours of rehydration via Gastrointestinal Symptom Rating Scale (GSRS).

Perceptual Data (6 per trial, maximal 9 minutes):

Thirst, stomach fullness, and taste, assessed via a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally physically active: Training > 2x per week and ≤ 6hours per week
* BMI of 18.5-29.9
* Stable weight for the last 2 months (<5 pounds. fluctuation)

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the trial
* night shifting work
* thyroid medication
* bariatric surgery
* cardiovascular disease
* renal disease
* hepatic disease
* Participating in another study at the same time
* Bodyweight <110 pounds
* Currently Smoker
* Major surgery, including abdominal, in the past 3 months or individuals who have planned surgery during the trial.
* Alcohol or drug abuse within the last 12 months
* High alcohol intake (average of > 2 standard drinks per day or > 10 standard drinks per week)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Net Fluid Balance | at 60 minutes, 120 minutes, 180 minutes and 240 minutes of rehydration
  Body water Retention after exercise-induced dehydration
Urine volume | 1, 2, 3, and 4 hour of the rehydration period
  Urine volume during the rehydration period
Free water clearance | 1, 2, 3, and 4 hours of the rehydration period
  Free water clearance during the rehydration period
Osmotic Clearance | 1, 2, 3, and 4 hours of the rehydration period
  Osmotic renal clearance during the rehydration period
Skin Hydration | 1, 2, 3, and 4 hours of the rehydration period
  Skin hydration at the face assessed with a moisture meter.

SECONDARY OUTCOMES:
Plasma Volume | 1, 2, 3, and 4 hours of the rehydration period
  Changes in Plasma Volume during rehydration based on hematocrit and hemoglobin
Stomach fullness | 1, 2, 3, and 4 hours of the rehydration period
  Stomach fullness assessed during dehydration
Gastrointestinal symptoms | At the end of the 4 hours rehydration period
  Gastrointestinal symptoms assessed with the structured assessment of gastrointestinal symptoms scale
Plasma Osmolality | 1, 2, 3, and 4 hours of the rehydration period
  Plasma osmolality during rehydration

CONTACTS AND LOCATIONS:
Locations (1):
- Hydration Science Lab, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided